CLINICAL TRIAL: NCT04567576
Title: Predictive Factors for COVID-19 in Rheumatology Study Based on Information Collected in The COVID-19 Global Rheumatology Alliance
Brief Title: Predictive Factors for COVID-19 in Rheumatology
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundación Santa Fe de Bogota (Other)
Responsible Party: Principal Investigator, Kevin Maldonado Cañón, Research Assistant, Fundación Santa Fe de Bogota
Other Study IDs: FPColCOVIDReuma2020
Record Dates: First submitted 2020-09-24; First posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Rheumatic Diseases; Covid19
MeSH Terms: conditions — Rheumatic Diseases; COVID-19 | interventions — Antirheumatic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed: Patients with underlying rheumatological or autoimmune diseases who have a confirmed infection by 2019-nCoV (COVID-19) who at the time of diagnosis (of infection) receive pharmacological treatment with disease modifying antirheumatic drugs (DMARDs).
  Interventions: Drug: Disease-modifying antirheumatic drugs (DMARDs)
- Un-exposed: Patients with underlying rheumatological or autoimmune diseases who have a confirmed 2019-nCoV (COVID-19) infection who at the time of diagnosis (of infection) are not receiving pharmacological treatment with disease-modifying antirheumatic drugs (DMARDs).

INTERVENTIONS:
Drug: Disease-modifying antirheumatic drugs (DMARDs) — Within a non-experimental setting, the routine disease-modifying antirheumatic drugs (DMARDs) prescription will be evaluated as the "exposure".
  Groups: Exposed

SUMMARY:
We seek to study the behaviour of Coronavirus infection in patients with rheumatological and/or autoimmune comorbidities, understood as a particular pathophysiological universe with its own risks and eventual benefits, until now fully hypothetical to be confirmed by means of real and recent evidence. On March 12, 2020, an initiative called the Global Alliance for COVID-19 in Rheumatology (The COVID-19 Rheumatology Alliance) arises, as a rapid response of international coordination whose ultimate goal is to serve as help or guideline for all those doctors who seek be faced with receiving, evaluating, understanding and caring for a patient with rheumatological and / or autoimmune diseases in relation to the imminent risk of COVID-19.

DETAILED DESCRIPTION:
Within this context, this study seeks to use the information registered by the Fundación Santa Fe de Bogotá University Hospital as a participating centre. It is intended, under a prospective cohort methodology, to identify, analyze and compare predictive factors of the clinical course of COVID-19 in patients with baseline diagnoses of rheumatological or autoimmune diseases with the intention of establishing well-founded parameters that contribute to the improvement in terms of strategies of prevention, management and prognosis; benefiting both directly treating physicians and patients, as well as indirectly a health system that is predicted to be pushed to the limit as time passes.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years.
* Have a diagnosis of a rheumatological disease and / or an autoimmune disease by meeting its own and standardized classification criteria.
* Confirmed diagnosis of COVID-19 by RT-PCR test
* Being a patient at the Fundación Santa Fe de Bogotá University Hospital.
* Be enroled in the registry of the Global Alliance for COVID-19 in Rheumatology.

Exclusion Criteria:

• Loss of follow-up due to referral to an institution other than the Fundación Santa Fe de Bogotá University Hospital, before documenting the outcome of his clinical picture.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have a confirmed or suspected COVID-19 infection and have been treated at the Santa Fe de Bogotá University Hospital.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Clinical behavior of the disease // COVID-19 | 1-12 weeks
  It will be considered as 1. Severe, if it meets at least one of the following characteristics (based on what is registered in the main center's database):
  * If you were hospitalized: What was the highest level of care you required during the illness? →
    o Required invasive mechanical ventilation or extracorporeal membrane oxygenation
  * If the symptoms did not resolve and the patient was hospitalized: What is the highest level of care that has been required in the course of the present illness so far? o Required mechanical ventilation or extracorporeal membrane oxygenation
Mortality | 1-12 weeks
  It will be considered as 1. Yes, if it meets at least one of the following characteristics (based on what is registered in the main center's database):
  • Has the patient died?
  o Yes, he passed away

IPD SHARING:
Plan to Share IPD: No